CLINICAL TRIAL: NCT05249231
Title: Parental Satisfaction of Hall Technique Versus Silver Diamine Fluoride (SDF) in the Management of Carious Primary Molars Randomized Clinical Trial
Brief Title: Parental Satisfaction of Hall Technique Versus SDF in the Management of Carious Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadir Emad, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6393
Record Dates: First submitted 2021-12-31; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Caries
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hall technique (Active Comparator): group of carious primary molars to be treated by hall technique
  Interventions: Device: Hall technique
- silver diamine fluoride (Experimental): group of carious primary molars to be treated by silver diamine fluoride
  Interventions: Drug: Silver diamine fluoride

INTERVENTIONS:
Drug: Silver diamine fluoride — Previous studies have recommended silver diamine fluoride (SDF) to exert a preventive result in managing early childhood caries ECC. However, no well-designed clinical trials have yet been performed to study the effect of SDF on caries prevention. The result is useful in arresting early childhood caries (ECC)
  Other Names: SDF
  Arms: silver diamine fluoride
Device: Hall technique — The first report on the Hall Technique published in 2007 by a general dental practitioner from Aberdeen/Scotland, Dr. Norna Hall. Dr. Hall used PMCs to restore carious primary molars rather than using the standard technique, placed them using a simplified method
  Other Names: HT
  Arms: Hall technique

SUMMARY:
* The aim of this study is to assess parental satisfaction and duration of the procedure of Hall and silver diamine fluoride techniques in the treatment of carious primary molars with healthy pulp.
* primary ourcome: parental satisfaction measurement device: four point likert scale measurement unit: 1-2-3-4
* secondary outcome: duration of the procedure measurement device: Digital chronometer measurement unit: minutes

DETAILED DESCRIPTION:
dental caries is a critical disease that affects primary teeth in early childhood. It occurs through interaction between acid-producing bacteria and carbohydrates on tooth surface. progression of caries depends on several factors such as type of diet, oral hygiene, cariogenic bacterial load and salivary flow. to control caries, the life style of a child should be improved by having healthy non-cariogenic diet and proper oral hygiene.

caries can be treated by advanced non-invasive methods such as: Hall technique and Silver diamine fluoride which are based on controlling the acidic medium of a cariogenic biofilm without removal of caries thus, arresting the progression of demineralization and restoring the function of diseased molars.

The first report on Hall Technique published in 2007 by a general dental practitioner from Aberdeen/Scotland, Dr. Norna Hall. Dr. Hall used PMCs to restore carious primary molars rather than using the standard technique through a more simplified method.

Previous studies have recommended silver diamine fluoride (SDF) to arrest early childhood caries ECC. However, no well-designed clinical trials have yet been performed to study the effect of SDF on caries prevention.

The trial is seeking the measurement of effectiveness of two modalities (Hall & SDF techniques) to achieve best acceptable treatment for caries in developing countries which have high caries index.

ELIGIBILITY:
Inclusion Criteria:

* 1 age: from 4 to 6 years old
* 2 primary molars with enamel/dentin caries without pulp exposure

Exclusion Criteria:

* 1 signs and symptoms of necrosis
* 2 root caries
* 3 spontaneous pain

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
parental satisfaction of Hall technique versus silver diamine fluoride | during procedure
  To estimate parental satisfaction with treatment, parents are going to be asked, "What's the level of your satisfaction with the treatment your child received? "Using a 4 point likert scale (very low equals 1, low equals 2, medium equals 3 and high equals 4)

SECONDARY OUTCOMES:
treatment time | during procedure
  Time will be measured from the start of the procedure till its end using digital chronometer as a device and minutes as a unit.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif B Eltaweil, prof, Study Director — Cairo University

REFERENCES:
- [Result] Ebrahimi M, Shirazi AS, Afshari E. Success and Behavior During Atraumatic Restorative Treatment, the Hall Technique, and the Stainless Steel Crown Technique for Primary Molar Teeth. Pediatr Dent. 2020 May 15;42(3):187-192. PMID 32522320
- See also: success and behavior during atraumatic restorative treatment, the hall technique and the stainless steel crown technique for primary molar teeth — http://pubmed.ncbi.nlm.nih.gov/32522320/